CLINICAL TRIAL: NCT07080892
Title: The Effect of Distal Versus Proximal Approach to the Interspace Between the Popliteal Artery and the Posterior Capsule of the Knee (iPACK) on Pain After Total Knee Arthroplasty
Brief Title: The Effect of Distal Versus Proximal iPACK on Pain After Total Knee Arthroplasty
Acronym: eDIPACK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNB/RU/052025
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain Following Knee Arthroplasty
Keywords: pain; postoperative pain; arthroplasty; peripheral nerve block; iPACK
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proximal iPACK group (Experimental): In the proximal iPACK group, participants will receive 20 ml of 0.25% levobupivacaine with adrenaline (1:200,000), injected at the level of the distal femoral shaft (a straight portion of the femur without the condyles).
  Interventions: Procedure: proximal iPACK
- distal iPACK group (Experimental): In the distal iPACK group, the participants will receive 20 ml of 0.25% levobupivacaine with adrenaline (1:200,000), injected at the most distal part of the thigh, between the femoral condyles.
  Interventions: Procedure: distal iPACK

INTERVENTIONS:
Procedure: distal iPACK — ● In the distal iPACK group, participants will receive 20 ml of 0.25% levobupivacaine with adrenaline (1:200,000), injected at the most distal part of the thigh, between the femoral condyles.
  Arms: distal iPACK group
Procedure: proximal iPACK — ● In the proximal iPACK group, participants will receive 20 ml of 0.25% levobupivacaine with adrenaline (1:200,000), injected at the level of the distal femoral shaft (a straight portion of the femur without the condyles).
  Arms: proximal iPACK group

SUMMARY:
Total knee arthroplasty (TKA) often results in significant postoperative pain, which can hinder recovery despite advances in surgical and anesthetic techniques. Traditional pain management methods like femoral nerve blocks may impair motor function, delaying rehabilitation. The iPACK block, targeting the posterior knee without affecting motor control, offers a promising alternative. This study aims to compare the effectiveness of two iPACK block approaches-proximal (at the distal femoral shaft) and distal (between the femoral condyles)-in managing postoperative pain in TKA patients. In a double-blind, randomized controlled trial with 120 participants, pain scores, opioid use, and time to rescue analgesia will be assessed. The hypothesis is that the distal iPACK block provides superior pain relief, potentially improving patient outcomes and recovery.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most frequently performed orthopedic procedures in modern medicine. Despite advancements in surgical techniques and perioperative care, postoperative pain management remains a significant challenge and a key factor influencing time to mobilization, patient satisfaction, and length of hospital stay. Commonly used analgesic techniques, such as femoral nerve blocks or epidural analgesia, while effective, can impair motor function and thus delay rehabilitation.

To minimize motor deficits while still providing effective pain relief, newer regional anesthesia techniques have been introduced into clinical practice. One such technique is the iPACK block (interspace between the popliteal artery and posterior capsule of the knee), which targets the posterior knee - an area often insufficiently covered by conventional nerve blocks. This method involves administering a local anesthetic into the space between the popliteal artery and the posterior capsule of the knee joint, offering analgesia without significant motor impairment.

Originally, the iPACK block was described as being performed at the level of the distal femoral shaft, several centimeters above the femoral condyles. Recently, however, a more distal variation of the technique has emerged, where the anesthetic is injected directly between the femoral condyles. This may provide more effective coverage of the posterior knee capsule's innervation. To date, there are no randomized trials that directly compare the efficacy of the distal and proximal iPACK approaches in terms of postoperative pain as the primary outcome.

Our aim is to conduct a prospective, randomized, placebo-controlled, double-blind clinical trial to compare the effectiveness of the distal and proximal iPACK blocks in patients undergoing TKA. A total of 120 patients will be enrolled and randomly assigned to one of two groups.

* In the proximal iPACK group, participants will receive 20 ml of 0.25% levobupivacaine with adrenaline (1:200,000), injected at the level of the distal femoral shaft (a straight portion of the femur without the condyles).
* In the distal iPACK group, the same volume and concentration of anesthetic will be injected at the most distal part of the thigh, between the femoral condyles.

All participants, regardless of group assignment, will also receive an adductor canal block with 20 ml of 0.25% levobupivacaine without adrenaline. In addition, all patients will receive standard analgesic therapy consisting of paracetamol (1 g IV every 8 hours) and diclofenac (75 mg IV every 12 hours). If necessary, rescue opioid doses will be available according to individual needs.

The efficacy of each approach will be assessed using several parameters: total opioid consumption within 24 hours and time to first opioid rescue dose, Visual Analogue Scale (VAS) both at rest and during active knee movement (up to 45 degrees) at 6, 12, and 24 hours postoperatively.

The hypothesis of our study is that the distal iPACK approach will provide more effective postoperative pain control compared to the original proximal technique. If confirmed, the findings could influence perioperative pain management protocols for TKA, support the broader adoption of the distal iPACK block in clinical practice, enhance patient comfort, reduce opioid use, promote earlier mobilization, and potentially shorten hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Patients undergoing primary unilateral total knee arthroplasty (TKA) for osteoarthritis
* Ability to understand and sign informed consent
* American Society of Anesthesiologists (ASA) classification I-III
* Ability to cooperate and participate in postoperative pain assessments (e.g., VAS)

Exclusion Criteria:

* Refusal to participate or failure to sign informed consent
* Bilateral or revision TKA
* Partial or unicondylar knee replacement
* Severe knee deformity (flexion, varus, or valgus >30°)
* Diagnosis other than osteoarthritis (e.g., rheumatoid arthritis, septic arthritis, post-traumatic arthritis)
* Allergy to local anesthetics or any medications used in the study
* Contraindications to regional anesthesia (e.g., infection at the injection site, coagulopathy, therapeutic anticoagulation)
* BMI > 40 kg/m²
* Severe renal impairment (KDIGO stage G4 or higher) or liver failure (Child-Pugh score ≥ 10)
* Prior surgery or vascular procedure on the femoral vessels of the operated limb
* Language barrier or inability to assess pain using the VAS
* Planned outpatient (same-day discharge) procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
total opioids consumption | from surgery until 24 hours after surgery
  total opioids consumption calculated to MME (morphine milligrams equivalent)

SECONDARY OUTCOMES:
time to first opioid administration | up to 24 hours after surgery
  time to first opioid administration time in hours to first opioid administration after operation.
Visual analog scale 6 (rest) | 6 hours postoperatively
  pain intensity will be measured using the Visual Analogue Scale at rest 6 hours postoperatively. The Visual Analogue Scale is a validated, 100-mm horizontal line used to measure pain intensity, ranging from "no pain" (0 mm) to "worst possible pain" (100 mm).
Visual analog scale 12 (rest) | 12 hours postoperatively
  pain intensity will be measured using the Visual Analogue Scale at rest 12 hours postoperatively. The Visual Analogue Scale is a validated, 100-mm horizontal line used to measure pain intensity, ranging from "no pain" (0 mm) to "worst possible pain" (100 mm).
Visual analog scale 24 (rest) | 24 hours postoperatively
  pain intensity will be measured using the Visual Analogue Scale at rest 24 hours postoperatively, The Visual Analogue Scale is a validated, 100-mm horizontal line used to measure pain intensity, ranging from "no pain" (0 mm) to "worst possible pain" (100 mm).
Visual analog scale 6 (flexion) | 6 hours postoperatively
  pain intensity will be measured using the Visual Analogue Scale at 45° flexion in the knee 6 hours postoperatively. The Visual Analogue Scale is a validated, 100-mm horizontal line used to measure pain intensity, ranging from "no pain" (0 mm) to "worst possible pain" (100 mm).
Visual analog scale 12 (flexion) | 12 hours postoperatively
  pain intensity will be measured using the Visual Analogue Scale at 45° flexion in the knee 12 hours postoperatively. The Visual Analogue Scale is a validated, 100-mm horizontal line used to measure pain intensity, ranging from "no pain" (0 mm) to "worst possible pain" (100 mm).
Visual analog scale 24 (flexion) | 24 hours postoperatively
  pain intensity will be measured using the Visual Analogue Scale at 45° flexion in the knee 24 hours postoperatively. The Visual Analogue Scale is a validated, 100-mm horizontal line used to measure pain intensity, ranging from "no pain" (0 mm) to "worst possible pain" (100 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Department of Anaesthesiology and Intensive Care Medicine, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No